CLINICAL TRIAL: NCT02952924
Title: A Safety, Tolerability, Pharmacokinetics and Efficacy Study of ro7049389 in: (1) Single- (With or Without Food) and Multiple- (With Midazolam) Ascending Doses in Healthy Volunteers; (2) Patients Chronically Infected With Hepatitis b Virus (3) Patients With Chronic Hepatitis B.
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of RO7049389 in Healthy Volunteers and Chronic Hepatitis B Virus (HBV) Infected Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YP39364
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- Parts 1a and 1b: SAD in Healthy Volunteers (Placebo) (Placebo Comparator): In Part 1a, participants will receive a single oral dose of placebo matching to RO7049389 film coated tablet on Day 1. In Part 1b, minimum 8 participants from Part 1a will be selected and 2 of whom will receive another single dose of placebo matching to RO7049389 on Day 16 after eating the standard United States - Food and Drug Administration (US FDA)-recommended high-fat and high-calorie breakfast.
  Interventions: Other: Placebo
- Parts 1a and 1b: SAD in Healthy Volunteers (RO7049389) (Experimental): In Part 1a, participants will receive a single oral dose of RO7049389 film coated tablet on Day 1 in dose-escalation cohorts with a starting dose of 150 milligrams (mg). The doses for subsequent cohorts will be defined by an adaptive approach based on the safety and PK data in previously-dosed healthy volunteers. In Part 1b, minimum 8 participants from Part 1a will be selected and 6 of whom will receive another single dose of RO7049389 on Day 16 after eating the standard US FDA-recommended high-fat and high-calorie breakfast.
  Interventions: Drug: RO7049389
- Part 1c: MAD in Healthy Volunteers (Placebo) (Placebo Comparator): Participants will receive placebo matching to RO7049389 film coated tablet from Days 1 to 13 (either once a day [QD] or twice a day [BID]) and a single dose of placebo matching to RO7049389 film coated tablet in the morning of Day 14. Participants will also receive a single dose of midazolam solution (100 micrograms [mcg]) on Day -1 and Day 14.
  Interventions: Drug: Midazolam; Other: Placebo
- Part 1c: MAD in Healthy Volunteers (RO7049389) (Experimental): Participants will receive RO7049389 film coated tablet from Days 1 to 13 (either QD or BID; dose and regimen will be decided based on the available PK and safety data) and a single dose of RO7049389 film coated tablet in the morning of Day 14. Participants will also receive a single dose of midazolam solution (100 mcg) on Day -1 and Day 14.
  Interventions: Drug: Midazolam; Drug: RO7049389
- Part 2: POM in Chronic HBV Participants (Placebo) (Placebo Comparator): Participants will receive placebo matching to RO7049389 film coated tablet from Days 1 to 27 (either QD or BID) and a single dose of placebo matching to RO7049389 film coated tablet in the morning of Day 28.
  Interventions: Other: Placebo
- Part 2: POM in Chronic HBV Participants (RO7049389) (Experimental): Participants will receive RO7049389 film coated tablet from Days 1 to 27 (either QD or BID; dose and regimen will be decided based on the available PK and safety data) and a single dose of RO7049389 film coated tablet in the morning of Day 28.
  Interventions: Drug: RO7049389
- Part 3: POM in NUC-Suppressed CHB Participants (Cohort A) (Experimental): Participants will receive RO7049389 on top of a NUC for 48 weeks at a dose determined from Part 2. NUC therapy will be administered per local label or guidelines.
  Interventions: Drug: RO7049389
- Part 3: POM in Treatment-Naive CHB Participants (Cohort B) (Experimental): Participants will receive RO7049389 for 4 weeks, followed by RO7049389 with an added NUC for 44 weeks. RO7049389 will be administered at a dose determined from Part 2. NUC therapy will be administered per local label or guidelines.
  Interventions: Drug: RO7049389
- Part 3: POM in Treatment-Naive CHB Participants (Cohort C) (Experimental): Participants will receive RO7049389 + NUC + Pegylated-Interferon (Peg-IFN) for 48 weeks. RO7049389 will be administered at a dose determined from Part 2. NUC and Peg-IFN therapy will be administered per local label or guidelines.
  Interventions: Drug: RO7049389

INTERVENTIONS:
Drug: Midazolam — Single dose of 100 mcg midazolam solution will be administered orally, before (Day -1) and after (Day 14) the treatment with RO7049389 or matching placebo
  Arms: Part 1c: MAD in Healthy Volunteers (Placebo); Part 1c: MAD in Healthy Volunteers (RO7049389)
Other: Placebo — Placebo matching to RO7049389 will be administered as per schedule described in individual arm.
  Arms: Part 1c: MAD in Healthy Volunteers (Placebo); Part 2: POM in Chronic HBV Participants (Placebo); Parts 1a and 1b: SAD in Healthy Volunteers (Placebo)
Drug: RO7049389 — RO7049389 will be administered as per schedule described in individual arm.
  Arms: Part 1c: MAD in Healthy Volunteers (RO7049389); Part 2: POM in Chronic HBV Participants (RO7049389); Part 3: POM in NUC-Suppressed CHB Participants (Cohort A); Part 3: POM in Treatment-Naive CHB Participants (Cohort B); Part 3: POM in Treatment-Naive CHB Participants (Cohort C); Parts 1a and 1b: SAD in Healthy Volunteers (RO7049389)

SUMMARY:
This study is a multicenter, three-part study. Parts 1 and 2 are randomized, investigator- and participant-blinded, placebo-control, single-ascending dose (SAD) and multiple-ascending dose (MAD) study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of RO7049389 following oral administration in healthy volunteers and chronic HBV infected participants. Part 3 is a non-randomized, non-controlled, open-label part to assess the efficacy and safety of RO7049389 when administered in combination with standard-of-care therapies for up to 48 weeks in nucleos(t)ide (NUC)-suppressed and treatment-naive chronic hepatitis B (CHB) participants.

ELIGIBILITY:
Inclusion Criteria:

Part 1- Healthy Volunteers only:

* Absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead Electrocardiogram (ECG), hematology, blood chemistry, serology and urinalysis
* A Body Mass Index (BMI) between 18 to 30 kilograms per square meter (kg/m^2) inclusive
* Female participants must be either surgically sterile or post-menopausal for at least one year
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Part 2- Chronic HBV-infected participants only:

* A BMI between 18 to 30 kg/m^2 inclusive
* Chronic Hepatitis B infection, defined as positive test for Hepatitis B surface antigen (HBsAg) for more than 6 months prior to randomization
* HBV DNA at screening greater than or equal to (>/=) 2 × 10^4 international units per milliliter (IU/mL) for Hepatitis B e antigen (HBeAg) positive participants, or >/=2 × 10^3 IU/mL for HBeAg-negative participants
* Liver biopsy, fibroscan or equivalent test obtained within the past 6 months demonstrating liver disease consistent with chronic HBV infection with absence of extensive bridging fibrosis and absence of cirrhosis
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm
* For women of childbearing potential: agreement to remain abstinent or use non-hormonal contraceptive methods that result in a failure rate of less than (<)1 percent (%) per year during the treatment period and for at least 3 months after the last dose of study drug

Part 3- Chronic HBV Participants Only:

* A BMI between 18 to 32 kg/m^2 inclusive
* Chronic hepatitis B infection, defined as positive test for HBsAg or HBV DNA, or positive HBeAg, for more than 6 months prior to screening
* For Cohorts only enrolling NUC-suppressed CHB participants (e.g. POM Cohort A), participants must have been treated with a single NUC (entecavir, tenofovir alafenamide, or tenofovir disoproxil fumarate) for at least 12 months. Participants must be on the same NUC therapy for at least 3 months prior to screening
* For Cohorts only enrolling anti-HBV treatment-naive and immune-active participants (e.g. POM Cohort B and Cohort C), previous anti-HBV treatments <30 days in total, and did not receive any anti-HBV treatments within 3 months prior to the first study dose
* Liver biopsy, fibroscan, or equivalent test obtained within the past 6 months demonstrating liver disease consistent with chronic HBV infection with absence of extensive bridging fibrosis and absence of cirrhosis
* For men: agreement to remain abstinent or use contraceptive measures, and agree to refrain from donating sperm
* For women of childbearing potential: agreement to remain abstinent or to use two approved contraceptive methods during the study and for at least 6 months after the last dose of study drug

Exclusion Criteria:

Part 1- Healthy Volunteers only:

* History or symptoms of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis
* History of Gilbert's syndrome
* Participants who have had significant acute infection, e.g., influenza, local infection, acute gastrointestinal symptoms or any other clinically significant illness within two weeks of dose administration
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies
* Any clinically significant concomitant diseases or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study
* Positive test at screening of any of the following: Hepatitis A (HAV IgM Ab), Hepatitis B (HBsAg), Hepatitis C (HCV RNA or HCV Ab) or human immunodeficiency virus (HIV Ab)
* Acute narrow-angle glaucoma (for MAD-midazolam cohorts)

Part 2- Chronic HBV-infected participants only:

* History or other evidence of bleeding from esophageal varices
* Evidence of liver cirrhosis or decompensated liver disease such as ascites, esophageal or gastric varices, splenomegaly, nodular liver, jaundice, hepatic encephalopathy
* History or other evidence of a medical condition associated with chronic liver disease other than HBV infection (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure, thalassemia, nonalcoholic steatohepatitis, etc.)
* Documented history or other evidence of metabolic liver disease within one year of randomization
* Positive test for hepatitis A (IgM anti-HAV), hepatitis C, hepatitis D, or human immunodeficiency virus
* History of or suspicion of hepatocellular carcinoma or alphafetoprotein >/= Upper limit of normal (ULN) at screening
* History of clinically significant gastrointestinal, cardiovascular, endocrine, renal, ocular, pulmonary, psychiatric or neurological disease
* History of organ transplantation
* Previous or concurrent HBV treatments in the past 6 months
* Significant acute infection (e.g., influenza, local infection) or any other clinically significant illness within 2 weeks of randomization

Part 3- Chronic Hepatitis B Participants Only:

* History or other evidence of bleeding from esophageal varices
* Evidence of liver cirrhosis or decompensated liver disease such as ascites, esophageal or gastric varices, splenomegaly, nodular liver, jaundice, or hepatic encephalopathy
* History or other evidence of a medical condition associated with chronic liver disease other than HBV infection (e.g. hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure, thalassemia, nonalcoholic statohepatitis, etc.)
* History of thyroid disease poorly controlled on prescribed medications or clinically relevant abnormal thyroid function tests
* Documented history or other evidence of metabolic liver disease within one year of screening
* Positive test for hepatitis A (IgM anti-HAV), hepatitis C, hepatitis D, HEV, or HIV
* Diagnosed or suspected hepatocellular carcinoma
* History of clinically significant gastrointestinal, cardiovascular, endocrine, renal, ocular, pulmonary, psychiatric, or neurological disease
* History of organ transplantation
* Significant acute infection (e.g. influenza, local infection) or any other clinically significant illness within 2 weeks of screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Melbourne Hospital, Parkville, Victoria
- Acibadem City Clinic Tokuda Hospital Ead, Sofia, Bulgaria
- China (3):
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
- Hong Kong (2):
  - The University of Hong Kong; Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- New Zealand (2):
  - Middlemore Hospital, Auckland
  - Auckland Clinical Studies Limited, Grafton
- Singapore (2):
  - National University Health System, Singapore
  - Singapore General Hospital, Singapore
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - Taichung Veterans Gen Hosp, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taipei
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai

REFERENCES:
- [Derived] Yuen MF, Zhou X, Gane E, Schwabe C, Tanwandee T, Feng S, Jin Y, Triyatni M, Lemenuel-Diot A, Cosson V, Xue Z, Kazma R, Bo Q. Safety, pharmacokinetics, and antiviral activity of RO7049389, a core protein allosteric modulator, in patients with chronic hepatitis B virus infection: a multicentre, randomised, placebo-controlled, phase 1 trial. Lancet Gastroenterol Hepatol. 2021 Sep;6(9):723-732. doi: 10.1016/S2468-1253(21)00176-X. Epub 2021 Jul 6. PMID 34237271
- [Derived] Feng S, Gane E, Schwabe C, Zhu M, Triyatni M, Zhou J, Bo Q, Jin Y. A Five-in-One First-in-Human Study To Assess Safety, Tolerability, and Pharmacokinetics of RO7049389, an Inhibitor of Hepatitis B Virus Capsid Assembly, after Single and Multiple Ascending Doses in Healthy Participants. Antimicrob Agents Chemother. 2020 Oct 20;64(11):e01323-20. doi: 10.1128/AAC.01323-20. Print 2020 Oct 20. PMID 32839221

RESULTS

PARTICIPANT FLOW:
Groups:
- Parts 1a and 1b: Single Ascending Dose (SAD) Placebo: Healthy volunteers (HVs) received a single dose of placebo under fasted (Part 1a) or fed (Part 1b) conditions.
- Part 1c: Multiple Ascending Dose (MAD) Placebo: HVs received placebo either once-daily (QD) or twice-daily (BID) for 13 days, followed by a single dose on Day 14.
- Part 2: Proof-of-Mechanism (POM) Placebo: Participants with chronic hepatitis B virus (CHB) infection received placebo once daily (QD) or twice daily (BID) for 27 days, followed by a single dose on Day 28.
- Part 1a: SAD Cohort 1: HVs received a single dose of 150 mg of RO7049389 under fasted conditions.
- Part 1a and Part 1b: SAD Cohort 2 (Food Effect): Part 1a: Single oral dose of 450 mg of RO7049389 under fasted conditions. Part 1b: Single oral dose of 450 mg of RO7049389 on Day 16 after a standard US FDA-recommended high-fat high-calorie meal.
- Part 1a: SAD Cohort 3; Part 1a: SAD Cohort 5: HVs received a single dose of 1000 mg of RO7049389 under fasted conditions.
- Part 1a: SAD Cohort 4: HVs received a single dose of 2000 mg of RO7049389 under fasted conditions.
- Part 1a: SAD Cohort 6: HVs received a single dose of 2500 mg of RO7049389 under fasted conditions.
- Part 1c: MAD Cohort 1: HVs received 200 mg of RO7049389 BID under fasted conditions for 13 days, followed by a single dose on Day 14. Participants also received a single oral dose of midazolam on Day -1 and Day 14.
- Part 1c: MAD Cohort 2: HVs received 200 mg of RO7049389 BID after a standard US FDA-recommended high-fat high-calorie meal for 13 days, followed by a single dose on Day 14. Participants also received a single oral dose of midazolam on Day -1 and Day 14.
- Part 1c: MAD Cohort 3: HVs received 400 mg of RO7049389 BID after a standard US FDA-recommended high-fat high-calorie meal for 13 days, followed by a single dose on Day 14. Participants also received a single oral dose of midazolam on Day -1 and Day 14.
- Part 1c: MAD Cohort 4: HVs received 800 mg of RO7049389 BID after a standard US FDA-recommended high-fat high-calorie meal for 13 days, followed by a single dose on Day 14. Participants also received a single oral dose of midazolam on Day -1 and Day 14.
- Part 1c: MAD Cohort 5: HVs received 600 mg of RO7049389 BID after a standard US FDA-recommended high-fat high-calorie meal for 13 days, followed by a single dose on Day 14. Participants also received a single oral dose of midazolam on Day -1 and Day 14.
- Part 2: POM Cohort 1: Participants with CHB received 200 mg of RO7049389 BID for 27 days after a standard US FDA recommended high-fat high-calorie meal, followed by a single dose on Day 28.
- Part 2: POM Cohort 2: Participants with CHB received 400 mg of RO7049389 BID for 27 days after a standard US FDA recommended high-fat high-calorie meal, followed by a single dose on Day 28.
- Part 2: POM Cohort 3: Participants with CHB received 600 mg of RO7049389 QD for 27 days under fasted conditions, followed by a single dose on Day 28.
- Part 2: POM Cohort 4: Participants with CHB received 1000 mg of RO7049389 QD for 27 days under fasted conditions, followed by a single dose on Day 28.
- Part 2: POM Cohort 5: Participants with CHB received 200 mg of RO7049389 QD for 27 days under fasted conditions, followed by a single dose on Day 28.
- Part 3: Cohort A: Nucleos(t)ide (NUC)-suppressed CHB participants received 600 mg of RO7049389 QD under fasted conditions in addition to an NUC (administered per local SoC) for 48 weeks. After the study treatment period, participants either continued NUC for another 24 weeks, or discontinued all treatment.
- Part 3: Cohort B: Treatment-naïve immune-active CHB participants 600 mg of RO7049389 QD under fasted conditions for 4 weeks, followed by RO7049389 + NUC (administered per local SoC) for an additional 44 weeks. After the study treatment period, participants either continued NUC for another 24 weeks, or discontinued all treatment.
- Part 3: Cohort C: Treatment-naïve immune-active CHB participants received 600 mg of RO7049389 QD under fasted conditions + NUC + pegylated interferon (Peg-IFN) for 48 weeks. After the study treatment period, participants either continued NUC for another 24 weeks, or discontinued all treatment.
Period: Overall Study
Arm/Group | Parts 1a and 1b: Single Ascending Dose (SAD) Placebo | Part 1c: Multiple Ascending Dose (MAD) Placebo | Part 2: Proof-of-Mechanism (POM) Placebo | Part 1a: SAD Cohort 1 | Part 1a and Part 1b: SAD Cohort 2 (Food Effect) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6 | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5 | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5 | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Started | 11 | 10 | 6 | 3 | 6 | 3 | 6 | 6 | 6 | 6 | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 32 | 10 | 30
Completed | 11 | 10 | 6 | 3 | 6 | 3 | 6 | 6 | 6 | 6 | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 31 | 10 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant refused to adhere to study protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant unable to adhere to study visit schedule | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Noncompliance with study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parts 1a and 1b: Single Ascending Dose (SAD) Placebo | Part 1c: Multiple Ascending Dose (MAD) Placebo | Part 2: Proof-of-Mechanism (POM) Placebo | Part 1a: SAD Cohort 1 | Part 1a and Part 1b: SAD Cohort 2 (Food Effect) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6 | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5 | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5 | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C | Total
Number analyzed (Participants) | 11 | 10 | 6 | 3 | 6 | 3 | 6 | 6 | 6 | 6 | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 32 | 10 | 30 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (8.4) | 25.2 (4.9) | 43.5 (6.4) | 32.7 (10.1) | 27.3 (7.6) | 28.7 (13.6) | 26.7 (4.7) | 26.7 (13.5) | 30.5 (7.0) | 25.5 (4.5) | 23.9 (2.8) | 26.7 (3.8) | 28.8 (11.1) | 28.3 (5.8) | 40.2 (8.3) | 34.7 (12.1) | 41.5 (11.8) | 47.0 (6.1) | 40.7 (15.3) | 47.2 (8.3) | 43.8 (9.8) | 32.8 (7.7) | 34.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 1 | 13 | 5 | 7 | 40
  Male | 10 | 10 | 3 | 3 | 6 | 3 | 6 | 6 | 6 | 6 | 7 | 7 | 6 | 6 | 5 | 3 | 4 | 3 | 5 | 19 | 5 | 23 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
  Not Hispanic or Latino | 10 | 8 | 6 | 3 | 6 | 2 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 7 | 6 | 30 | 9 | 30 | 180
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 5 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 3 | 1 | 1 | 5 | 5 | 5 | 7 | 5 | 25 | 5 | 28 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 10
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 9 | 7 | 0 | 1 | 5 | 3 | 6 | 3 | 6 | 4 | 7 | 4 | 3 | 4 | 1 | 0 | 1 | 0 | 1 | 6 | 4 | 1 | 76
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Adverse Events
Time Frame: Up to Day 29 (Part 1a), Day 44 (Part 1b), Day 42 (Part 1c)
Population: The safety analysis population included all participants who received at least one dose of study drug, whether prematurely withdrawn from the study or not.
Measure: Number; unit: Percentage of participants
Arm/Group | Parts 1a and 1b: Single Ascending Dose (SAD) Placebo | Part 1a: SAD Cohort 1 | Part 1a and Part 1b: SAD Cohort 2 (Food Effect) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6 | Part 1c: Multiple Ascending Dose (MAD) Placebo | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 11 | 3 | 6 | 3 | 6 | 6 | 6 | 10 | 6 | 7 | 7 | 6 | 6
Percentage of participants | 27.3 | 33.3 | 50.0 | 100 | 83.3 | 33.3 | 50.0 | 60.0 | 83.3 | 57.1 | 28.6 | 16.7 | 16.7

2. Primary Outcome: Parts 1a and 1b: SAD Cohort: Time to Reach Maximum Concentration (Tmax) of RO7049389
Time Frame: Up to 28 days
Population: The pharmacokinetic population included all participants unless they significantly violated inclusion/exclusion criteria, deviated significantly from the protocol, or if they had unavailable or incomplete data that could affect analysis.
Measure: Median (Full Range); unit: Hours
Groups:
- Part 1a : SAD Cohort 2 (Food Effect - Fasted): Part 1a: Single oral dose of 450 mg of RO7049389 under fasted conditions.
- Part 1b: SAD Cohort 2 (Food Effect - Fed): Part 1b: Single oral dose of 450 mg of RO7049389 on Day 16 after a standard US FDA-recommended high-fat high-calorie meal.
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a : SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6 | 6 | 6
Hours | 2.0 [2.0 to 2.0] | 1.25 [1.0 to 2.0] | 3.0 [1.5 to 4.0] | 1.5 [1.5 to 3.0] | 2.0 [1.5 to 3.0] | 1.5 [1.5 to 3.0] | 3.0 [1.5 to 4.0]

3. Primary Outcome: Parts 1a and 1b: SAD Cohort: Maximum Observed Plasma Concentration (Cmax) of RO7049389
Time Frame: Up to 28 days
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a : SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6 | 6 | 6
ng/mL | 250 (33.4) | 1900 (79.7) | 4610 (75.6) | 8990 (77.4) | 14700 (67.6) | 8990 (77.4) | 24800 (63.9)

4. Primary Outcome: Parts 1a and 1b: SAD Cohort: AUC From Time Zero to Infinity (AUC0-inf) of RO7049389
Time Frame: Up to 28 days
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a : SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6 | 6 | 6
ng*hr/mL | 879 (7.5) | 4690 (53.2) | 10900 (71.9) | 34400 (71.6) | 46300 (62.0) | 34400 (71.6) | 134000 (91.4)

5. Primary Outcome: Parts 1a and 1b: SAD Cohort: Area Under the Curve From Time Zero to the Last Measurable Concentration (AUC0-last) of RO7049389
Time Frame: Up to 28 days
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a : SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6 | 6 | 6
ng*hr/mL | 868 (6.6) | 4660 (53.8) | 10900 (72.0) | 34300 (71.6) | 46200 (62.1) | 34300 (71.6) | 134000 (91.4)

6. Primary Outcome: Parts 1a and 1b: SAD Cohort: Half-life (T1/2) of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a : SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6 | 6 | 6
Hours | 3.34 (35.3) | 8.80 (81.1) | 4.20 (32.0) | 7.23 (39.5) | 12.1 (52.1) | 7.23 (39.5) | 12.4 (44.7)

7. Primary Outcome: Parts 1a and 1b: SAD Cohort: Apparent Oral Clearance (CL/F) of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a : SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6 | 6 | 6
L/hr | 171 (7.3) | 128 (67.8) | 61.5 (72.1) | 64.9 (130.3) | 63.3 (69.7) | 64.9 (130.3) | 69.7 (122.3)

8. Primary Outcome: Parts 1a and 1b: SAD Cohort: Cumulative Amount Excreted Unchanged in Urine (Ae) of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a : SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 0 | 6 | 0 | 3 | 6 | 6 | 6
mg |  | 0.312 (69.6) |  | 1.88 (83.9) | 3.56 (92.0) | 1.88 (83.9) | 6.89 (101.8)

9. Primary Outcome: Parts 1a and 1b: SAD Cohort: Renal Clearance (CLr) of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Groups:
- Part 1a: SAD Cohort 2 (Food Effect - Fasted): Part 1a: Single oral dose of 450 mg of RO7049389 under fasted conditions.
Arm/Group | Part 1a: SAD Cohort 1 | Part 1a: SAD Cohort 2 (Food Effect - Fasted) | Part 1b: SAD Cohort 2 (Food Effect - Fed) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6
Number analyzed (Participants) | 0 | 6 | 0 | 3 | 6 | 6 | 6
mL/min |  | 1.60 (84.8) |  | 1.55 (42.9) | 1.41 (18.7) | 1.55 (42.9) | 0.82 (22.8)

10. Primary Outcome: Part 2: Percentage of Participants With Adverse Events
Time Frame: Up to Day 112
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Proof-of-Mechanism (POM) Placebo | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6
Percentage of participants | 50.0 | 66.7 | 66.7 | 83.3 | 57.1 | 33.3

11. Primary Outcome: Part 2: Quantitative Plasma HBV DNA Level
Time Frame: Baseline - Day 112
Population: The efficacy population included all participants who received at least one dose of RO7049389.
Measure: Median (Full Range); unit: Log10 IU/mL
Arm/Group | Part 2: Proof-of-Mechanism (POM) Placebo | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6
Log10 IU/mL
  Baseline | 5.94 [4.8 to 8.2] | 4.50 [1.9 to 8.3] | 7.80 [4.0 to 8.5] | 4.43 [3.3 to 8.4] | 5.10 [4.1 to 8.7] | 7.14 [3.9 to 8.5]
  Day 8: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6
  Day 8 | 5.25 [4.6 to 7.8] | 1.40 [1.3 to 4.8] | 5.27 [1.8 to 6.2] | 1.75 [1.3 to 5.7] | 2.25 [1.3 to 6.5] | 5.21 [2.0 to 6.0]
  Day 15: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 15 | 5.29 [4.3 to 8.1] | 2.00 [1.3 to 5.4] | 4.58 [1.4 to 6.0] | 1.46 [1.3 to 5.5] | 1.30 [1.3 to 6.0] | 4.90 [1.3 to 5.6]
  Day 22: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 22 | 5.16 [3.8 to 8.0] | 1.83 [1.3 to 5.1] | 4.11 [1.3 to 5.8] | 1.41 [1.3 to 5.2] | 1.41 [1.3 to 5.6] | 4.65 [1.3 to 5.4]
  Day 28: number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6
  Day 28 | 5.29 [3.6 to 8.0] | 1.65 [1.3 to 4.9] | 3.64 [1.3 to 5.8] | 1.30 [1.3 to 4.9] | 1.30 [1.3 to 5.5] | 4.43 [1.3 to 5.4]
  Day 35/Follow-up Day 7: number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6
  Day 35/Follow-up Day 7 | 5.29 [2.7 to 8.0] | 3.23 [1.3 to 8.0] | 5.50 [2.8 to 6.6] | 2.61 [1.5 to 6.9] | 2.98 [2.4 to 6.7] | 6.29 [2.4 to 7.6]
  Day 56/Follow-up Day 28: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 56/Follow-up Day 28 | 5.21 [2.7 to 8.1] | 4.07 [2.4 to 8.3] | 6.53 [3.3 to 8.2] | 3.43 [2.8 to 9.1] | 4.04 [3.1 to 8.3] | 7.07 [3.9 to 8.3]
  Day 84/Follow-up Day 56: number analyzed (Participants) | 5 | 4 | 5 | 6 | 6 | 6
  Day 84/Follow-up Day 56 | 5.15 [2.6 to 8.2] | 5.76 [2.4 to 8.0] | 5.68 [4.4 to 8.1] | 4.29 [3.5 to 8.2] | 4.73 [3.7 to 8.5] | 6.83 [3.8 to 8.4]
  Day 112/Follow-up Day 84: number analyzed (Participants) | 5 | 4 | 6 | 6 | 6 | 6
  Day 112/Follow-up Day 84 | 5.09 [3.0 to 8.0] | 5.89 [3.2 to 7.9] | 6.17 [4.1 to 8.2] | 4.45 [3.2 to 8.4] | 4.55 [4.0 to 8.4] | 7.03 [3.8 to 8.3]

12. Primary Outcome: Part 3: Proportion of Patients Achieving Functional Cure
Description: Functional cure is defined as HBV DNA < lower limit of quantification (LLOQ, 20 IU/mL) with HBsAg loss (< 0.05 IU/mL) at 24 weeks post-treatment.
Time Frame: Every 2-4 weeks from Baseline through Week 72
Population: The ITT population included all participants who were randomized and received at least one dose of study drug (RO7049389 or placebo). Participants were analyzed according to the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Percentage
  Baseline | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 2 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 4 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 8 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 12 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 16 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 20 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 24 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 28 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 32 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 36 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 40 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 44 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 48 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 50 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 52 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 54 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 56 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 58 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 60 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 64 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 68 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]
  Week 72 | 0 [0 to 0.11] | 0 [0 to 0.31] | 0 [0 to 0.12]

13. Secondary Outcome: Part 1b: Food Effect on Cmax of RO7049389
Description: This outcome measure evaluated the effect of food on the pharmacokinetics (PK) of RO7049389 after the administration of a single dose. Participants were fed a high-fat, high-calorie breakfast (per FDA food effect bioavailability and bioequivalence study recommendations) 30 minutes prior to dosing after fasting overnight for at least 8 hours. ANOVA (factors fasted/fed state and subject) was performed for measurements available in subjects in both fasted and fed states.
Time Frame: Day 16
Measure: Geometric Mean (90% Confidence Interval); unit: geometric mean ratio
Arm/Group | Part 1a and Part 1b: SAD Cohort 2 (Food Effect)
Number analyzed (Participants) | 6
geometric mean ratio | 2.42 [1.48 to 3.95]

14. Secondary Outcome: Part 1b: Food Effect on AUCinf of RO7049389
Description: as for outcome 13
Time Frame: Day 16
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: geometric mean ratio
Arm/Group | Part 1a and Part 1b: SAD Cohort 2 (Food Effect)
Number analyzed (Participants) | 6
geometric mean ratio | 2.17 [1.39 to 3.40]

15. Secondary Outcome: Part 1c: Cmax of Midazolam
Description: This endpoint presents the geometric mean ratio (after RO7049389/before RO7049389).
Time Frame: Up to Day 14
Population: The pharmacokinetic population included all participants unless they significantly violated inclusion/exclusion criteria, deviated significantly from the protocol, or if they had unavailable or incomplete data that could affect analysis. Cohort 4 was terminated after 3 days of administration and could not be included in analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 6 | 6
Ratio | 0.892 [0.663 to 1.20] | 1.01 [0.846 to 1.21] | 1.12 [0.915 to 1.37] | 0.940 [0.734 to 1.21]

16. Secondary Outcome: Part 1c: AUCinf of Midazolam
Description: This endpoint presents the geometric mean ratio (after RO7049389/before RO7049389).
Time Frame: Up to Day 14
Population: as for outcome 15
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio | 1.10 [0.846 to 1.42] | 1.18 [1.06 to 1.31] | 1.25 [1.04 to 1.50] | 1.16 [0.993 to 1.36]

17. Secondary Outcome: Part 1c: Tmax of RO7049389
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
hours
  Day 1 | 2.0 [1.5 to 3.0] | 2.0 [1.5 to 3.0] | 3.0 [1.5 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 3.0]
  Day 14: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6
  Day 14 | 1.5 [1.0 to 1.5] | 2.0 [1.5 to 4.0] | 3.0 [1.5 to 4.0] |  | 3.0 [3.0 to 4.0]

18. Secondary Outcome: Part 1c: Cmax of RO7049389
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
ng/mL
  Day 1 | 483 (42.5) | 840 (41.7) | 4840 (53.7) | 14500 (39.5) | 10600 (42.2)
  Day 14: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6
  Day 14 | 735 (19.9) | 583 (41.3) | 2720 (49.0) |  | 9960 (32.7)

19. Secondary Outcome: Part 1c: AUC0-12hr of RO7049389
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
ng*hr/mL
  Day 1 | 1304.09 (31.9) | 1819.92 (46.1) | 9760.31 (55.7) | 32459.87 (42.6) | 27041.94 (33.6)
  Day 14: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6
  Day 14 | 1806.59 (25.6) | 1573.32 (27.5) | 6511.21 (29.0) |  | 28051.71 (32.5)

20. Secondary Outcome: Part 1c: CLr of RO7049389
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
mL/min
  Day 1 | 1.06 (74.2) | 1.08 (82.6) | 1.43 (27.0) | 2.04 (54.7) | 1.19 (48.6)
  Day 14: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6
  Day 14 | 1.96 (75.2) | 1.87 (51.7) | 3.01 (46.9) |  | 2.32 (35.0)

21. Secondary Outcome: Part 1c: Accumulation Ratio of RO7049389
Description: This endpoint presents the geometric mean ratio of AUC after a single dose (Day 1) and AUC after having received multiple doses (Day 14) within each arm.
Time Frame: Day 1, Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Geometric mean ratio
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6
Geometric mean ratio | 1.45 (24.3) | 1.05 (31.1) | 0.880 (35.6) | 1.09 (37.4)

22. Secondary Outcome: Part 1c: T1/2 of RO7049389
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
Hours
  Day 1 | 2.27 (24.1) | 2.44 (12.6) | 2.09 (18.5) | 1.70 (30.4) | 1.53 (22.5)
  Day 14: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6
  Day 14 | 5.79 (40.7) | 5.17 (26.8) | 5.08 (10.5) |  | 5.73 (28.9)

23. Secondary Outcome: Part 1c: Ae of RO7049389
Time Frame: Up to Day 14
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
mg
  Day 1 | 0.0926 (90.7) | 0.0900 (56.0) | 0.859 (60.9) | 3.58 (63.4) | 1.77 (35.9)
  Day 14: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6
  Day 14 | 0.243 (89.5) | 0.189 (60.7) | 1.26 (53.8) |  | 3.68 (26.3)

24. Secondary Outcome: Part 1c: Ctrough of RO7049389
Time Frame: Up to Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6
ng/mL | 12.1 (45.1) | 15.2 (27.8) | 42.1 (12.8) | 88.9 (27.6)

25. Secondary Outcome: Part 2: HBV DNA < Lower Limit of Quantification (LLOQ)
Time Frame: Baseline - Day 112/Follow-up Day 84
Population: The efficacy population included all participants who received at least one dose of RO7049389.
Measure: Number; unit: Percentage of participants
Groups:
- Part 2: POM Placebo: Participants with chronic hepatitis B virus (CHB) infection received placebo once daily (QD) or twice daily (BID) for 27 days, followed by a single dose on Day 28.
Arm/Group | Part 2: POM Placebo | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6
Percentage of participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6
  Day 8 | 0 | 33.3 | 0 | 50.0 | 28.6 | 0
  Day 15: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 15 | 0 | 50.0 | 0 | 50.0 | 57.1 | 16.7
  Day 22: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 22 | 0 | 50.0 | 0 | 50.0 | 42.9 | 16.7
  Day 28: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 28 | 0 | 50.0 | 16.7 | 66.7 | 57.1 | 16.7
  Day 35/Follow-up Day 7: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 35/Follow-up Day 7 | 0 | 16.7 | 0 | 0 | 0 | 0
  Day 56/Follow-up Day 28: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
  Day 56/Follow-up Day 28 | 0 | 0 | 0 | 0 | 0 | 0
  Day 84/Follow-up Day 56: number analyzed (Participants) | 5 | 4 | 5 | 6 | 6 | 6
  Day 84/Follow-up Day 56 | 0 | 0 | 0 | 0 | 0 | 0
  Day 112/Follow-up Day 84: number analyzed (Participants) | 5 | 4 | 6 | 6 | 6 | 6
  Day 112/Follow-up Day 84 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Part 2: Tmax of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
Hours
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 1 | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0] | 1.97 [0.92 to 3.0] | 1.98 [1.92 to 3.03] | 1.5 [1.0 to 2.87]
  Day 28: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 28 | 2.5 [1.08 to 3.0] | 2.5 [2.0 to 4.0] | 2.0 [0.97 to 3.0] | 2.03 [1.90 to 2.85] | 1.5 [0.833 to 3.0]

27. Secondary Outcome: Part 2: Cmax of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
ng/mL
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 1 | 1450 (69.1) | 8110 (59.7) | 5030 (42.7) | 23900 (41.8) | 910 (89.1)
  Day 28: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 28 | 1500 (60.3) | 8580 (63.7) | 4890 (76.9) | 29800 (15.2) | 998 (52.8)

28. Secondary Outcome: Part 2: AUCtau of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
ng*hr/mL
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 1 | 2870 (50.2) | 19900 (78.6) | 11500 (65.5) | 80000 (71.2) | 3500 (76.7)
  Day 28: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 28 | 3350 (47.7) | 22400 (70.5) | 14600 (78.0) | 133000 (50.0) | 3480 (56.9)

29. Secondary Outcome: Part 2: Accumulation Ratio of RO7049389
Description: This endpoint presents the geometric mean ratio of AUC after a single dose (Day 1) and AUC after having received multiple doses (Day 28) within each arm.
Time Frame: Day 1, Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Geometric mean ratio
Arm/Group | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Geometric mean ratio | 1.01 (81.3) | 0.971 (58.2) | 1.65 (109.8) | 0.823 (77.0) | 0.917 (40.9)

30. Secondary Outcome: Part 2: T1/2 of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
Hours
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 1 | 1.68 (18.0) | 1.15 (27.6) | 1.09 (22.4) | 1.40 (34.5) | 2.33 (55.2)
  Day 28: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Day 28 | 3.38 (24.1) | 3.26 (28.8) | 3.70 (26.1) | 2.33 (20.1) | 3.81 (24.6)

31. Secondary Outcome: Part 2: Ctrough of RO7049389
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 26.7 (72.7) | 68.2 (89.2) | 7.94 (60.6) | 27.0 (42.3) | 3.37 (88.1)

32. Secondary Outcome: Part 3: Percentage of Participants With AEs
Time Frame: 72 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Percentage of Participants | 68.8 | 90 | 100

33. Secondary Outcome: Part 3: Hepatitis B Surface Antigen (HBsAg) Level
Time Frame: Baseline - Week 72
Population: as for outcome 12
Measure: Median (Full Range); unit: Log10 IU/mL
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Log10 IU/mL
  Baseline | 3.04 [2.48 to 4.30] | 3.51 [2.44 to 4.63] | 4.10 [2.50 to 5.49]
  Week 2: number analyzed (Participants) | 31 | 10 | 29
  Week 2 | 3.08 [2.42 to 4.36] | 3.51 [2.53 to 4.69] | 4.14 [2.18 to 5.63]
  Week 4: number analyzed (Participants) | 31 | 10 | 30
  Week 4 | 3.08 [2.52 to 4.33] | 3.47 [2.36 to 4.46] | 3.98 [1.74 to 5.55]
  Week 8: number analyzed (Participants) | 30 | 10 | 29
  Week 8 | 3.00 [2.41 to 4.33] | 3.49 [2.30 to 4.25] | 3.62 [1.34 to 5.06]
  Week 12: number analyzed (Participants) | 30 | 10 | 30
  Week 12 | 3.02 [2.42 to 4.31] | 3.52 [2.51 to 4.25] | 3.55 [1.44 to 4.82]
  Week 16: number analyzed (Participants) | 30 | 9 | 29
  Week 16 | 3.03 [2.59 to 4.28] | 3.22 [2.64 to 4.25] | 3.44 [1.56 to 4.46]
  Week 20: number analyzed (Participants) | 30 | 10 | 29
  Week 20 | 3.05 [2.54 to 4.30] | 3.48 [2.79 to 4.26] | 3.26 [1.47 to 4.37]
  Week 24: number analyzed (Participants) | 30 | 9 | 29
  Week 24 | 2.99 [2.58 to 4.25] | 3.84 [2.85 to 4.23] | 3.15 [0.98 to 4.30]
  Week 28: number analyzed (Participants) | 30 | 10 | 29
  Week 28 | 3.04 [2.58 to 4.27] | 3.39 [2.81 to 4.29] | 3.10 [1.04 to 4.33]
  Week 32: number analyzed (Participants) | 30 | 8 | 29
  Week 32 | 2.99 [2.54 to 4.28] | 3.52 [3.12 to 4.32] | 3.09 [0.82 to 4.27]
  Week 36: number analyzed (Participants) | 30 | 10 | 28
  Week 36 | 2.98 [2.47 to 4.32] | 3.50 [2.85 to 4.20] | 2.93 [0.83 to 4.21]
  Week 40: number analyzed (Participants) | 30 | 9 | 28
  Week 40 | 3.03 [2.52 to 4.26] | 3.81 [2.80 to 4.21] | 2.91 [0.80 to 4.24]
  Week 44: number analyzed (Participants) | 30 | 9 | 28
  Week 44 | 3.00 [2.50 to 4.23] | 3.81 [2.84 to 4.24] | 2.91 [0.38 to 4.20]
  Week 48: number analyzed (Participants) | 30 | 10 | 28
  Week 48 | 2.99 [2.50 to 4.23] | 3.53 [2.81 to 4.18] | 2.90 [0.05 to 4.15]
  Week 50: number analyzed (Participants) | 11 | 2 | 5
  Week 50 | 2.96 [2.55 to 4.21] | 3.21 [3.18 to 3.24] | 0.83 [0.21 to 1.72]
  Week 52: number analyzed (Participants) | 10 | 2 | 5
  Week 52 | 2.89 [2.55 to 4.24] | 3.21 [3.20 to 3.23] | 1.32 [0.37 to 1.78]
  Week 54: number analyzed (Participants) | 9 | 4 | 5
  Week 54 | 2.98 [2.53 to 4.29] | 3.51 [3.16 to 3.89] | 1.41 [0.36 to 2.02]
  Week 56: number analyzed (Participants) | 30 | 9 | 28
  Week 56 | 2.97 [2.48 to 4.21] | 3.75 [2.82 to 4.20] | 2.86 [0.45 to 4.25]
  Week 58: number analyzed (Participants) | 3 | 1 | 5
  Week 58 | 2.67 [2.52 to 4.23] | 3.15 [3.15 to 3.15] | 1.70 [0.48 to 2.19]
  Week 60: number analyzed (Participants) | 6 | 2 | 5
  Week 60 | 3.84 [2.52 to 4.22] | 3.20 [3.16 to 3.23] | 1.79 [0.50 to 2.25]
  Week 64: number analyzed (Participants) | 31 | 8 | 28
  Week 64 | 2.98 [2.50 to 4.23] | 3.53 [2.85 to 4.00] | 2.83 [0.76 to 4.85]
  Week 68: number analyzed (Participants) | 2 | 1 | 5
  Week 68 | 2.65 [2.56 to 2.74] | 3.12 [3.12 to 3.12] | 1.84 [1.00 to 2.46]
  Week 72: number analyzed (Participants) | 31 | 9 | 28
  Week 72 | 2.95 [2.49 to 4.17] | 3.71 [2.83 to 4.23] | 2.75 [0.78 to 4.30]

34. Secondary Outcome: Part 3: Hepatitis B e-Antigen (HBeAg) Levels
Time Frame: Baseline - Week 72
Population: The population for this endpoint included participants in Part 3 that were HBeAg+ at baseline.
Measure: Median (Full Range); unit: Log10 IU/mL
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 11 | 6 | 19
Log10 IU/mL
  Baseline | 0.17 [-0.54 to 1.93] | 1.07 [0.00 to 2.44] | 2.84 [1.48 to 3.49]
  Week 2 | 0.16 [-0.54 to 2.31] | 1.01 [-0.89 to 2.31] | 2.79 [1.16 to 3.55]
  Week 4 | 0.17 [-0.54 to 2.01] | 0.60 [-0.89 to 1.96] | 2.57 [0.65 to 3.36]
  Week 8 | 0.15 [-0.54 to 1.78] | 0.33 [-0.89 to 1.19] | 2.24 [0.24 to 2.80]
  Week 12 | 0.12 [-0.54 to 1.74] | 0.17 [-0.89 to 0.57] | 2.02 [0.20 to 2.55]
  Week 16: number analyzed (Participants) | 11 | 6 | 18
  Week 16 | 0.12 [-0.54 to 1.71] | -0.04 [-0.89 to 0.39] | 1.81 [-0.24 to 2.36]
  Week 20: number analyzed (Participants) | 11 | 6 | 18
  Week 20 | 0.06 [-0.54 to 1.55] | -0.12 [-0.89 to 0.37] | 1.40 [-0.89 to 2.25]
  Week 24: number analyzed (Participants) | 11 | 6 | 18
  Week 24 | 0.10 [-0.54 to 1.38] | -0.24 [-0.89 to 0.38] | 1.31 [-0.89 to 2.10]
  Week 28: number analyzed (Participants) | 11 | 6 | 18
  Week 28 | 0.12 [-0.54 to 1.39] | -0.32 [-0.89 to 0.28] | 1.32 [-0.89 to 2.03]
  Week 32: number analyzed (Participants) | 11 | 6 | 18
  Week 32 | 0.14 [-0.54 to 1.14] | -0.40 [-0.89 to 0.38] | 1.12 [-0.89 to 1.97]
  Week 36: number analyzed (Participants) | 11 | 6 | 18
  Week 36 | 0.15 [-0.54 to 1.21] | -0.43 [-0.89 to 0.29] | 0.96 [-0.89 to 1.89]
  Week 40: number analyzed (Participants) | 11 | 5 | 18
  Week 40 | 0.13 [-0.54 to 1.16] | -0.49 [-0.89 to 0.21] | 0.83 [-0.89 to 1.82]
  Week 44: number analyzed (Participants) | 11 | 6 | 18
  Week 44 | 0.16 [-0.54 to 1.14] | -0.50 [-0.89 to 0.34] | 0.82 [-0.89 to 1.75]
  Week 48: number analyzed (Participants) | 11 | 6 | 18
  Week 48 | 0.15 [-0.54 to 1.16] | -0.52 [-0.89 to 0.20] | 0.69 [-0.89 to 1.79]
  Week 50: number analyzed (Participants) | 2 | 2 | 1
  Week 50 | -0.53 [-0.54 to -0.52] | -0.71 [-0.89 to -0.54] | -0.47 [-0.47 to -0.47]
  Week 52: number analyzed (Participants) | 2 | 2 | 1
  Week 52 | -0.54 [-0.54 to -0.54] | -0.71 [-0.89 to -0.54] | -0.54 [-0.54 to -0.54]
  Week 54: number analyzed (Participants) | 1 | 2 | 1
  Week 54 | -0.54 [-0.54 to -0.54] | -0.54 [-0.54 to -0.54] | -0.49 [-0.49 to -0.49]
  Week 56: number analyzed (Participants) | 11 | 6 | 18
  Week 56 | 0.09 [-0.54 to 1.22] | -0.54 [-0.89 to 0.22] | 0.74 [-0.89 to 2.08]
  Week 58: number analyzed (Participants) | 0 | 1 | 1
  Week 58 |  | -0.54 [-0.54 to -0.54] | 1.23 [1.23 to 1.23]
  Week 60: number analyzed (Participants) | 0 | 1 | 1
  Week 60 |  | -0.54 [-0.54 to -0.54] | 1.70 [1.70 to 1.70]
  Week 64: number analyzed (Participants) | 11 | 4 | 18
  Week 64 | 0.14 [-0.54 to 1.21] | -0.54 [-0.89 to -0.30] | 0.36 [-0.89 to 2.96]
  Week 68: number analyzed (Participants) | 0 | 1 | 1
  Week 68 |  | -0.54 [-0.54 to -0.54] | -0.54 [-0.54 to -0.54]
  Week 72: number analyzed (Participants) | 11 | 5 | 18
  Week 72 | 0.08 [-0.54 to 1.16] | -0.35 [-0.89 to 0.36] | -0.23 [-0.89 to 1.96]

35. Secondary Outcome: Part 3: HBV RNA Level
Time Frame: Baseline - Week 72
Population: as for outcome 12
Measure: Median (Full Range); unit: Log10 copies/mL
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Log10 copies/mL
  Baseline | 0.99 [0.69 to 4.45] | 4.02 [0.69 to 6.24] | 5.30 [0.69 to 7.50]
  Week 2: number analyzed (Participants) | 31 | 10 | 29
  Week 2 | 0.69 [0.69 to 1.79] | 1.04 [0.69 to 3.93] | 2.37 [0.69 to 4.53]
  Week 4: number analyzed (Participants) | 31 | 10 | 30
  Week 4 | 0.69 [0.69 to 1.35] | 0.84 [0.69 to 2.90] | 1.93 [0.69 to 4.97]
  Week 8: number analyzed (Participants) | 30 | 10 | 29
  Week 8 | 0.69 [0.69 to 2.45] | 0.69 [0.69 to 1.68] | 1.54 [0.69 to 7.03]
  Week 12: number analyzed (Participants) | 29 | 10 | 29
  Week 12 | 0.69 [0.69 to 2.64] | 0.69 [0.69 to 0.99] | 0.99 [0.69 to 3.37]
  Week 16: number analyzed (Participants) | 30 | 9 | 29
  Week 16 | 0.69 [0.69 to 1.65] | 0.69 [0.69 to 0.99] | 0.99 [0.69 to 3.08]
  Week 20: number analyzed (Participants) | 29 | 10 | 29
  Week 20 | 0.69 [0.69 to 0.99] | 0.69 [0.69 to 0.99] | 0.99 [0.69 to 3.24]
  Week 24: number analyzed (Participants) | 30 | 9 | 29
  Week 24 | 0.69 [0.69 to 0.99] | 0.69 [0.69 to 0.99] | 0.99 [0.69 to 3.09]
  Week 28: number analyzed (Participants) | 30 | 10 | 28
  Week 28 | 0.69 [0.69 to 0.99] | 0.69 [0.69 to 0.99] | 0.99 [0.69 to 3.03]
  Week 32: number analyzed (Participants) | 29 | 8 | 29
  Week 32 | 0.69 [0.69 to 0.99] | 0.69 [0.69 to 0.99] | 0.99 [0.69 to 2.87]
  Week 36: number analyzed (Participants) | 29 | 10 | 28
  Week 36 | 0.69 [0.69 to 1.22] | 0.69 [0.69 to 0.69] | 0.99 [0.69 to 2.92]
  Week 40: number analyzed (Participants) | 28 | 9 | 28
  Week 40 | 0.69 [0.69 to 1.89] | 0.69 [0.69 to 0.69] | 0.99 [0.69 to 2.65]
  Week 44: number analyzed (Participants) | 30 | 9 | 28
  Week 44 | 0.69 [0.69 to 0.99] | 0.69 [0.69 to 0.99] | 0.99 [0.69 to 2.73]
  Week 48: number analyzed (Participants) | 30 | 10 | 28
  Week 48 | 0.69 [0.69 to 1.83] | 0.69 [0.69 to 0.69] | 0.99 [0.69 to 2.70]
  Week 50: number analyzed (Participants) | 11 | 2 | 5
  Week 50 | 0.69 [0.69 to 1.48] | 1.02 [0.69 to 1.34] | 0.99 [0.69 to 0.99]
  Week 52: number analyzed (Participants) | 10 | 2 | 5
  Week 52 | 0.69 [0.69 to 1.75] | 1.46 [1.04 to 1.88] | 0.99 [0.69 to 0.99]
  Week 54: number analyzed (Participants) | 9 | 4 | 5
  Week 54 | 0.69 [0.69 to 1.64] | 2.08 [0.69 to 2.76] | 0.99 [0.69 to 0.99]
  Week 56: number analyzed (Participants) | 30 | 9 | 28
  Week 56 | 0.99 [0.69 to 4.07] | 1.94 [0.69 to 3.44] | 1.54 [0.69 to 6.09]
  Week 58: number analyzed (Participants) | 3 | 1 | 5
  Week 58 | 0.69 [0.69 to 1.44] | 1.75 [1.75 to 1.75] | 0.99 [0.69 to 2.49]
  Week 60: number analyzed (Participants) | 6 | 2 | 5
  Week 60 | 0.69 [0.69 to 1.89] | 1.25 [0.69 to 1.82] | 0.99 [0.69 to 2.65]
  Week 64: number analyzed (Participants) | 31 | 8 | 28
  Week 64 | 0.99 [0.69 to 3.85] | 1.28 [0.69 to 2.82] | 0.99 [0.69 to 5.98]
  Week 68: number analyzed (Participants) | 2 | 1 | 5
  Week 68 | 1.28 [0.99 to 1.56] | 1.99 [1.99 to 1.99] | 0.99 [0.99 to 1.10]
  Week 72: number analyzed (Participants) | 31 | 9 | 28
  Week 72 | 0.99 [0.69 to 3.87] | 1.77 [0.69 to 4.52] | 1.08 [0.69 to 6.04]

36. Secondary Outcome: Part 3: HBV Core-Related Antigen (HBcrAg) Levels
Time Frame: Baseline - Week 72
Population: as for outcome 12
Measure: Median (Full Range); unit: Log10 U/mL
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Log10 U/mL
  Baseline | 4.10 [1.90 to 6.90] | 6.15 [2.90 to 7.80] | 7.95 [1.90 to 9.10]
  Week 2: number analyzed (Participants) | 31 | 10 | 29
  Week 2 | 4.10 [1.90 to 6.80] | 5.95 [1.90 to 7.60] | 7.80 [1.90 to 9.00]
  Week 4: number analyzed (Participants) | 31 | 10 | 30
  Week 4 | 4.20 [1.90 to 6.80] | 5.55 [1.90 to 7.20] | 7.00 [1.90 to 8.70]
  Week 8: number analyzed (Participants) | 30 | 10 | 29
  Week 8 | 4.30 [1.90 to 6.80] | 5.25 [1.90 to 6.50] | 6.70 [1.90 to 8.90]
  Week 12: number analyzed (Participants) | 30 | 10 | 30
  Week 12 | 4.30 [1.90 to 6.70] | 5.15 [1.90 to 6.20] | 6.30 [1.90 to 8.80]
  Week 16: number analyzed (Participants) | 30 | 9 | 29
  Week 16 | 4.05 [1.90 to 6.60] | 5.50 [2.90 to 6.00] | 6.20 [2.50 to 8.70]
  Week 20: number analyzed (Participants) | 30 | 10 | 29
  Week 20 | 4.10 [2.50 to 6.70] | 5.00 [2.90 to 6.00] | 5.90 [2.50 to 8.30]
  Week 24: number analyzed (Participants) | 29 | 9 | 29
  Week 24 | 4.20 [2.90 to 6.60] | 5.10 [2.50 to 5.90] | 5.70 [1.90 to 8.00]
  Week 28: number analyzed (Participants) | 30 | 10 | 29
  Week 28 | 4.05 [2.50 to 6.40] | 5.00 [1.90 to 5.90] | 5.60 [2.50 to 7.70]
  Week 32: number analyzed (Participants) | 30 | 8 | 29
  Week 32 | 4.20 [2.50 to 6.50] | 4.85 [2.90 to 6.10] | 5.40 [1.90 to 9.10]
  Week 36: number analyzed (Participants) | 30 | 10 | 28
  Week 36 | 4.05 [2.90 to 6.40] | 5.10 [2.90 to 6.10] | 5.45 [1.90 to 7.80]
  Week 40: number analyzed (Participants) | 30 | 9 | 28
  Week 40 | 4.10 [2.90 to 6.50] | 4.90 [2.50 to 6.10] | 5.45 [2.50 to 7.50]
  Week 44: number analyzed (Participants) | 30 | 9 | 28
  Week 44 | 4.35 [2.90 to 6.40] | 4.80 [2.50 to 6.10] | 5.35 [1.90 to 7.80]
  Week 48: number analyzed (Participants) | 30 | 10 | 28
  Week 48 | 4.10 [2.50 to 6.60] | 5.10 [2.90 to 6.00] | 5.45 [2.50 to 9.10]
  Week 50: number analyzed (Participants) | 11 | 2 | 5
  Week 50 | 4.00 [1.90 to 4.80] | 5.05 [4.80 to 5.30] | 3.10 [2.90 to 4.80]
  Week 52: number analyzed (Participants) | 10 | 2 | 5
  Week 52 | 3.60 [1.90 to 4.90] | 5.05 [4.90 to 5.20] | 3.10 [2.90 to 4.80]
  Week 54: number analyzed (Participants) | 9 | 4 | 5
  Week 54 | 3.30 [2.50 to 4.80] | 3.90 [2.50 to 5.50] | 3.10 [2.90 to 4.90]
  Week 56: number analyzed (Participants) | 30 | 9 | 28
  Week 56 | 4.15 [2.50 to 6.50] | 5.00 [2.90 to 6.10] | 5.50 [1.90 to 9.10]
  Week 58: number analyzed (Participants) | 3 | 1 | 5
  Week 58 | 2.50 [2.50 to 4.60] | 5.30 [5.30 to 5.30] | 3.20 [2.90 to 6.10]
  Week 60: number analyzed (Participants) | 6 | 2 | 5
  Week 60 | 4.15 [2.50 to 4.70] | 3.60 [2.50 to 4.70] | 2.90 [2.50 to 6.50]
  Week 64: number analyzed (Participants) | 31 | 8 | 28
  Week 64 | 4.20 [2.50 to 6.50] | 4.40 [2.90 to 5.60] | 5.15 [1.90 to 9.10]
  Week 68: number analyzed (Participants) | 2 | 1 | 5
  Week 68 | 3.80 [2.90 to 4.70] | 5.30 [5.30 to 5.40] | 3.20 [3.00 to 4.40]
  Week 72: number analyzed (Participants) | 31 | 9 | 28
  Week 72 | 4.20 [1.90 to 6.40] | 4.80 [2.50 to 6.50] | 4.70 [1.90 to 9.10]

37. Secondary Outcome: Part 3: Alanine Transaminase (ALT) Normalization in Participants With Baseline ALT Elevation
Time Frame: Week 12 - Week 72
Population: This endpoint includes participants from Part 3 with elevated ALT at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 0 | 9 | 28
Percentage of participants
  Week 12 |  | 66.67 | 35.71
  Week 24 |  | 88.89 | 62.96
  Week 36 |  | 88.89 | 77.78
  Week 48 |  | 88.89 | 85.19
  Week 56 |  | 77.78 | 81.48
  Week 64 |  | 100 | 92.59
  Week 72 |  | 87.5 | 92.59

38. Secondary Outcome: Part 3: Percentage of Participants With Anti-Hepatitis B Core Antigen (HBc) Antibodies
Time Frame: Up to Week 72
Population: This endpoint included participants from Part 3 who were anti-HBc+ at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Percentage of participants | 100 | 100 | 100

39. Secondary Outcome: Part 3: HBV DNA Level
Time Frame: Baseline - Week 72
Population: as for outcome 12
Measure: Median (Full Range); unit: Log10 copies/mL
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Log10 copies/mL
  Baseline | 1.28 [1.28 to 1.28] | 6.06 [2.61 to 8.84] | 7.37 [3.43 to 9.36]
  Week 2: number analyzed (Participants) | 31 | 10 | 29
  Week 2 | 1.28 [1.28 to 1.28] | 3.14 [1.28 to 6.47] | 3.89 [0.95 to 6.40]
  Week 4: number analyzed (Participants) | 31 | 10 | 30
  Week 4 | 1.28 [1.28 to 1.28] | 1.99 [1.28 to 5.44] | 2.76 [0.95 to 5.78]
  Week 8: number analyzed (Participants) | 30 | 10 | 29
  Week 8 | 1.28 [1.28 to 1.28] | 1.41 [1.28 to 3.73] | 1.54 [0.95 to 6.15]
  Week 12: number analyzed (Participants) | 29 | 10 | 30
  Week 12 | 1.28 [1.28 to 1.91] | 1.28 [1.28 to 1.97] | 1.44 [0.95 to 4.69]
  Week 16: number analyzed (Participants) | 30 | 9 | 29
  Week 16 | 1.28 [1.28 to 1.41] | 1.28 [1.28 to 2.33] | 1.28 [0.95 to 3.99]
  Week 20: number analyzed (Participants) | 30 | 10 | 29
  Week 20 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 2.01] | 1.28 [0.95 to 3.28]
  Week 24: number analyzed (Participants) | 30 | 9 | 29
  Week 24 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.45] | 1.28 [0.95 to 2.55]
  Week 28: number analyzed (Participants) | 29 | 10 | 29
  Week 28 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.28] | 1.28 [0.95 to 2.55]
  Week 32: number analyzed (Participants) | 30 | 8 | 28
  Week 32 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.43] | 1.28 [0.95 to 4.11]
  Week 36: number analyzed (Participants) | 30 | 10 | 28
  Week 36 | 1.28 [1.28 to 1.32] | 1.28 [1.28 to 1.41] | 1.28 [0.95 to 2.21]
  Week 40: number analyzed (Participants) | 30 | 9 | 28
  Week 40 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.62] | 1.28 [0.95 to 2.08]
  Week 44: number analyzed (Participants) | 30 | 9 | 28
  Week 44 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.28] | 1.28 [0.95 to 2.39]
  Week 48: number analyzed (Participants) | 30 | 10 | 27
  Week 48 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.28] | 1.28 [0.95 to 2.10]
  Week 50: number analyzed (Participants) | 11 | 2 | 5
  Week 50 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.28] | 0.95 [0.95 to 1.28]
  Week 52: number analyzed (Participants) | 10 | 2 | 5
  Week 52 | 1.28 [1.28 to 1.59] | 1.28 [1.28 to 1.28] | 1.28 [0.95 to 2.01]
  Week 54: number analyzed (Participants) | 9 | 4 | 5
  Week 54 | 1.28 [1.28 to 1.30] | 1.28 [1.28 to 1.28] | 1.28 [0.95 to 2.89]
  Week 56: number analyzed (Participants) | 30 | 9 | 28
  Week 56 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.53] | 1.28 [0.95 to 5.02]
  Week 58: number analyzed (Participants) | 3 | 1 | 5
  Week 58 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.28] | 2.09 [0.95 to 4.88]
  Week 60: number analyzed (Participants) | 6 | 2 | 5
  Week 60 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.28] | 2.52 [0.95 to 5.23]
  Week 64: number analyzed (Participants) | 31 | 6 | 28
  Week 64 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 2.94] | 1.28 [0.95 to 6.65]
  Week 68: number analyzed (Participants) | 2 | 1 | 5
  Week 68 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 1.28] | 2.67 [0.95 to 4.66]
  Week 72: number analyzed (Participants) | 30 | 9 | 28
  Week 72 | 1.28 [1.28 to 1.28] | 1.28 [1.28 to 6.33] | 1.28 [0.95 to 4.70]

40. Secondary Outcome: Part 3: HBV DNA < Lower Limit of Quantification (LLOQ)
Time Frame: Baseline - Week 72
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Percentage of participants
  Baseline | 100 | 0 | 0
  Week 2: number analyzed (Participants) | 31 | 10 | 29
  Week 2 | 100 | 10 | 10.3
  Week 4: number analyzed (Participants) | 31 | 10 | 30
  Week 4 | 100 | 30 | 16.7
  Week 8: number analyzed (Participants) | 30 | 10 | 29
  Week 8 | 100 | 40 | 41.4
  Week 12: number analyzed (Participants) | 28 | 10 | 30
  Week 12 | 96.4 | 70 | 43.3
  Week 16: number analyzed (Participants) | 30 | 9 | 29
  Week 16 | 96.7 | 77.8 | 51.7
  Week 20: number analyzed (Participants) | 30 | 10 | 29
  Week 20 | 100 | 90 | 55.2
  Week 24: number analyzed (Participants) | 30 | 9 | 29
  Week 24 | 100 | 88.9 | 51.7
  Week 28: number analyzed (Participants) | 29 | 10 | 29
  Week 28 | 100 | 100 | 55.2
  Week 32: number analyzed (Participants) | 30 | 8 | 28
  Week 32 | 100 | 87.5 | 64.3
  Week 36: number analyzed (Participants) | 30 | 10 | 28
  Week 36 | 96.7 | 90 | 67.9
  Week 40: number analyzed (Participants) | 30 | 9 | 28
  Week 40 | 100 | 77.8 | 71.4
  Week 44: number analyzed (Participants) | 30 | 9 | 28
  Week 44 | 100 | 100 | 71.4
  Week 48: number analyzed (Participants) | 30 | 10 | 27
  Week 48 | 100 | 100 | 81.5
  Week 50: number analyzed (Participants) | 11 | 2 | 5
  Week 50 | 100 | 100 | 100
  Week 52: number analyzed (Participants) | 10 | 2 | 5
  Week 52 | 90 | 100 | 80
  Week 54: number analyzed (Participants) | 9 | 4 | 5
  Week 54 | 88.9 | 100 | 80
  Week 56: number analyzed (Participants) | 30 | 9 | 28
  Week 56 | 100 | 88.9 | 64.3
  Week 58: number analyzed (Participants) | 3 | 1 | 5
  Week 58 | 100 | 100 | 40
  Week 60: number analyzed (Participants) | 6 | 2 | 5
  Week 60 | 100 | 100 | 20
  Week 64: number analyzed (Participants) | 31 | 6 | 28
  Week 64 | 100 | 83.3 | 67.9
  Week 68: number analyzed (Participants) | 2 | 1 | 5
  Week 68 | 100 | 100 | 40
  Week 72: number analyzed (Participants) | 30 | 9 | 28
  Week 72 | 100 | 77.8 | 78.6

41. Secondary Outcome: Part 3: Tmax of RO7049389
Time Frame: Day 1 - Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Hours
  Day 1 | 1.99 [0.98 to 3.03] | 2.00 [1.00 to 3.02] | 1.96 [0.95 to 3.02]
  Week 4: number analyzed (Participants) | 0 | 9 | 0
  Week 4 |  | 2.02 [1.00 to 3.02] |
  Week 24: number analyzed (Participants) | 30 | 9 | 29
  Week 24 | 1.94 [0.00 to 3.00] | 2.00 [1.00 to 3.00] | 2.00 [0.92 to 4.15]
  Week 48: number analyzed (Participants) | 30 | 10 | 28
  Week 48 | 1.02 [0.00 to 3.13] | 2.50 [1.00 to 3.05] | 2.00 [0.93 to 3.97]

42. Secondary Outcome: Part 3: Cmax of RO7049389
Time Frame: Day 1 - Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
ng/mL
  Day 1 | 7140 (107.6) | 5390 (94.3) | 5910 (116.8)
  Week 4: number analyzed (Participants) | 0 | 9 | 0
  Week 4 |  | 4630 (92.8) |
  Week 24: number analyzed (Participants) | 30 | 9 | 30
  Week 24 | 2500 (2040.7) | 3900 (126.9) | 4260 (89.4)
  Week 48: number analyzed (Participants) | 30 | 10 | 30
  Week 48 | 5410 (88.4) | 3510 (246.1) | 3570 (133.6)

43. Secondary Outcome: Part 3: AUCtau of RO7049389
Time Frame: Day 1 - Week 48
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
h*ng/mL
  Day 1: number analyzed (Participants) | 32 | 8 | 25
  Day 1 | 18700 (105.1) | 16700 (79.3) | 20900 (107.4)
  Week 4: number analyzed (Participants) | 0 | 9 | 0
  Week 4 |  | 13600 (117.2) |
  Week 24: number analyzed (Participants) | 26 | 8 | 23
  Week 24 | 15400 (121.3) | 10500 (241.8) | 13200 (88.2)
  Week 48: number analyzed (Participants) | 28 | 8 | 27
  Week 48 | 14100 (84.8) | 16000 (121.3) | 11700 (107.6)

44. Secondary Outcome: Part 3: T1/2 of RO7049389
Time Frame: Day 1 - Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
Number analyzed (Participants) | 32 | 10 | 30
Hours
  Day 1: number analyzed (Participants) | 32 | 8 | 25
  Day 1 | 1.16 [0.757 to 1.67] | 1.13 [0.891 to 1.31] | 1.31 [0.899 to 1.98]
  Week 4: number analyzed (Participants) | 0 | 10 | 0
  Week 4 |  | 1.38 [0.897 to 1.89] |
  Week 24: number analyzed (Participants) | 26 | 8 | 23
  Week 24 | 1.30 [0.832 to 2.19] | 1.43 [1.17 to 2.38] | 1.38 [1.06 to 2.25]
  Week 48: number analyzed (Participants) | 27 | 8 | 27
  Week 48 | 4.05 [2.62 to 7.59] | 3.40 [2.63 to 5.85] | 3.98 [2.54 to 8.33]

ADVERSE EVENTS:
Time Frame: Up to Day 29 (Part 1a), Day 44 (Part 1b), Day 42 (Part 1c), Day 112 (Part 2), and 72 weeks (Part 3)
Arm/Group | Parts 1a and 1b: Single Ascending Dose (SAD) Placebo | Part 1c: Multiple Ascending Dose (MAD) Placebo | Part 2: Proof-of-Mechanism (POM) Placebo | Part 1a: SAD Cohort 1 | Part 1a and Part 1b: SAD Cohort 2 (Food Effect) | Part 1a: SAD Cohort 3 | Part 1a: SAD Cohort 4 | Part 1a: SAD Cohort 5 | Part 1a: SAD Cohort 6 | Part 1c: MAD Cohort 1 | Part 1c: MAD Cohort 2 | Part 1c: MAD Cohort 3 | Part 1c: MAD Cohort 4 | Part 1c: MAD Cohort 5 | Part 2: POM Cohort 1 | Part 2: POM Cohort 2 | Part 2: POM Cohort 3 | Part 2: POM Cohort 4 | Part 2: POM Cohort 5 | Part 3: Cohort A | Part 3: Cohort B | Part 3: Cohort C
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/6 | 0/3 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/32 | 1/10 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 1/6 | 0/3 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 1/32 | 1/10 | 2/30
Other Adverse Events (participants affected / at risk) | 3/11 | 6/10 | 3/6 | 1/3 | 3/6 | 3/3 | 5/6 | 2/6 | 3/6 | 5/6 | 4/7 | 2/7 | 1/6 | 1/6 | 4/6 | 4/6 | 5/6 | 4/7 | 2/6 | 22/32 | 9/10 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parts 1a and 1b: Single Ascending Dose (SAD) Placebo (N=11) | Part 1c: Multiple Ascending Dose (MAD) Placebo (N=10) | Part 2: Proof-of-Mechanism (POM) Placebo (N=6) | Part 1a: SAD Cohort 1 (N=3) | Part 1a and Part 1b: SAD Cohort 2 (Food Effect) (N=6) | Part 1a: SAD Cohort 3 (N=3) | Part 1a: SAD Cohort 4 (N=6) | Part 1a: SAD Cohort 5 (N=6) | Part 1a: SAD Cohort 6 (N=6) | Part 1c: MAD Cohort 1 (N=6) | Part 1c: MAD Cohort 2 (N=7) | Part 1c: MAD Cohort 3 (N=7) | Part 1c: MAD Cohort 4 (N=6) | Part 1c: MAD Cohort 5 (N=6) | Part 2: POM Cohort 1 (N=6) | Part 2: POM Cohort 2 (N=6) | Part 2: POM Cohort 3 (N=6) | Part 2: POM Cohort 4 (N=7) | Part 2: POM Cohort 5 (N=6) | Part 3: Cohort A (N=32) | Part 3: Cohort B (N=10) | Part 3: Cohort C (N=30)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parts 1a and 1b: Single Ascending Dose (SAD) Placebo (N=11) | Part 1c: Multiple Ascending Dose (MAD) Placebo (N=10) | Part 2: Proof-of-Mechanism (POM) Placebo (N=6) | Part 1a: SAD Cohort 1 (N=3) | Part 1a and Part 1b: SAD Cohort 2 (Food Effect) (N=6) | Part 1a: SAD Cohort 3 (N=3) | Part 1a: SAD Cohort 4 (N=6) | Part 1a: SAD Cohort 5 (N=6) | Part 1a: SAD Cohort 6 (N=6) | Part 1c: MAD Cohort 1 (N=6) | Part 1c: MAD Cohort 2 (N=7) | Part 1c: MAD Cohort 3 (N=7) | Part 1c: MAD Cohort 4 (N=6) | Part 1c: MAD Cohort 5 (N=6) | Part 2: POM Cohort 1 (N=6) | Part 2: POM Cohort 2 (N=6) | Part 2: POM Cohort 3 (N=6) | Part 2: POM Cohort 4 (N=7) | Part 2: POM Cohort 5 (N=6) | Part 3: Cohort A (N=32) | Part 3: Cohort B (N=10) | Part 3: Cohort C (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 1 (1) | 5 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (6)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (13)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 5 (9)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 18 (35)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Mumps (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 11 (13)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 9 (12)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (12)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (17)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (11)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (12)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (9)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (10)
Headache (Nervous system disorders) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (7) | 2 (3) | 14 (20)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (2) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 11 (11)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02952924/Prot_SAP_000.pdf